CLINICAL TRIAL: NCT01432613
Title: Diagnostic Accuracy of Whole Body Magnetic Resonance Imaging in Inflammatory Myopathies
Acronym: DARWIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K071204
Record Dates: First submitted 2011-08-22; First posted 2011-09-13 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Myositis; Polymyositis; Dermatomyositis; Myositis, Inclusion Body
Keywords: Myositis; Magnetic Resonance Imaging; Muscle biopsy; Sensitivity and Specificity
MeSH Terms: conditions — Myositis; Polymyositis; Dermatomyositis; Myositis, Inclusion Body; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI-oriented muscle biopsy (Other): Muscle sample will be done following the usual care.
  Interventions: Procedure: MRI-oriented muscle biopsy

INTERVENTIONS:
Procedure: MRI-oriented muscle biopsy — Orientation of muscle biopsy according to the MRI results

SUMMARY:
Idiopathic inflammatory myopathies (IIM) are a great concern in acquired muscle illnesses. An appropriate and rapid diagnosis is necessary, because morbidity and mortality are high and a specific treatment is needed. Currently the use of muscle MRI (magnetic resonance imaging) in departments managing IIM is common. In absence of recommendations fixing their place in the diagnostic phase, the practices observed are extremely heterogeneous. This practices diversity well reflects the lack of data in the literature, making it impossible to appreciate the real contribution of this test. The main aim of this interventional study is to evaluate the diagnostic accuracy of muscle MRI (in terms of sensitivity, specificity, predictive positive value and predictive negative value) for patients who are suspected to suffer from IIM.

DETAILED DESCRIPTION:
Idiopathic inflammatory myopathies (IIM) are a great concern in acquired muscle illnesses. An appropriate and rapid diagnosis is necessary, because morbidity and mortality are high and as a specific treatment is needed (corticosteroids, immunosuppressant, and "biotherapies").

Currently the use of muscle MRI in departments managing IIM is common. In absence of recommendations fixing their place in the diagnostic phase, the practices observed are extremely heterogeneous. Some systematically order a muscle MRI for patients suspected to suffer from IIM, others hold this examination for patients selected according to non defined criteria, and others sometimes use MRI to follow-up patients. This practices diversity well reflects the lack of data in the literature, making it impossible to appreciate the real contribution of this test. The results published in the great majority of studies are obtained with patients whose IIM diagnosis is already established. The diagnostic accuracy of muscle MRI in real conditions of clinical practice is thus unknown for patients having a simple suspicion of IIM.

Primary scientific aim: Evaluation of diagnostic accuracy of muscle MRI (in terms of sensitivity, specificity, predictive positive value and predictive negative value) for patients who are suspected to suffer from IIM.

Secondary scientific aim: Comparison of two diagnostic strategies: MRI-oriented muscle biopsy versus non MRI-oriented muscle biopsy.

Gold standard: muscle biopsy Index test: whole body MRI, STIR and T1 sequences Patients and setting of diagnosis tests: Screening will be realized on any patient suspected to suffer from inflammatory and addressed for muscle biopsy in one of the participating reference centres for neuro-muscular disorders. -Evaluate if RMI is efficiency to reduce false negative results during a second biopsy.

* Evaluation of reproducibility inter-observers and intra-observers of interpretations of RMI.
* Evaluation of reproducibility inter-observers and intra-observers of muscles biopsy interpretations according with the European neuro muscular classification ENMC.

Study calendar :

* Including 130 patients during 24 months
* RMI interpretations are realised immediately after RMI exam without informing the investigator.
* Procedures of anonymisation of the double reading are done every 03 months.

  * V1 = inclusion visit Information and non-opposition of patient Collection of demographic, clinical and biological data
  * V2 = muscle MRI
  * V3 = muscle biopsy
  * One year after V1, collection of the final established diagnosis and compare it to the investigator results

ELIGIBILITY:
Inclusion Criteria:

* Skin rash typical of dermatomyositis: "lilac" rash (+/- oedemata) of upper eyelids, periungual sign, erythematous-scaly eruption occurring over the MCP and IPP, elbow, knees (Gottron's signs ands papules), erythema of light-sensitive areas OR
* Muscle weakness which is proximal, bilateral and objectifiable by clinical examination ≤ 4/5, and CPK≥2N (N<170).
* Increase CPK and presence of acquired myositis specific antibody

AND

-Onset of troubles ≤3 years

Exclusion Criteria:

* Pregnant female
* Proximal motive neuropathy
* Refusing participation
* Patient under 18 years old
* Adult patient under legal protection
* Patient with contraindication for MRI, pacemaker
* For all other magnetic or ironic implanted equipments, metal workers, must contact PI to ensure their eligibility
* Ocular muscles weakness, isolated dysarthria,
* Patients suffering from toxic myopathy, amyloidosis, inherited muscular dystrophy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2010-12-22 (Actual); Primary Completion 2016-02-11 (Actual); Study Completion 2016-11-26 (Actual)

PRIMARY OUTCOMES:
Evaluation of T1 and STIR (Short Tau Inversion Recovery) sequences of muscle MRI. | between Day 0 and 24 months
  Description : diagnostic accuracy of muscle MRI (in terms of sensitivity, specificity, predictive positive value and predictive negative value) for the diagnostic of inflammatory myopathy.
Presence of IIM diagnosed by muscle biopsy | between Day 0 and 24 months
  Presence of IIM according to ENMC histological criteria

SECONDARY OUTCOMES:
Evaluation of reproductibility intra- versus inter-observers for muscle biopsy interpretation | every 3 months (up to 24 months)
  Evaluation of reproductibility intra- versus inter-observers for muscle biopsy interpretation according to ENMC (European Neuromuscular Centre) classification (calculation of Kappa coefficients).
Evaluation of reproductibility intra- versus inter-observers for muscle MRI interpretation | every 3 months (up to 24 months)
  Evaluation of reproductibility intra- versus inter-observers for muscle MRI interpretation (calculation of Kappa coefficients).

CONTACTS AND LOCATIONS:
Overall Officials: Yves ALLENBACH, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- CHU Amiens Nord, Amiens, France

IPD SHARING:
Plan to Share IPD: No